CLINICAL TRIAL: NCT04409015
Title: ROTEM® Obstetric Hemorrhage Pilot Study
Status: Completed | Type: Observational
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Michael Cackovic, MD, Associate Professor, Ohio State University
Other Study IDs: 2020H0119
Record Dates: First submitted 2020-05-26; First posted 2020-06-01 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: High Risk Postpartum Hemorrhage (PPH)
Keywords: High risk Postpartum hemorrhage (PPH); ROTEM; pregnant women

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: ROTEM - rotation thromboelastometry testing — The ROTEM® is a simple blood test that provides information about specific components involved in blood clotting and stopping hemorrhage.

SUMMARY:
This is a prospective observational study among women at high-risk of postpartum hemorrhage, in their third trimester who are admitted to Labor &Delivery in spontaneous labor, for induction of labor, or for scheduled cesarean section.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years and able to provide consent
2. Gestational age ≥ 34 weeks
3. ≥ 1 High-risk of postpartum hemorrhage criteria defined as either of:

   1. Nulliparous women admitted for induction of labor with unfavorable cervix (Bishop's score <5)
   2. Prior uterine surgery (> 1 prior cesarean or myomectomy)
   3. Patients undergoing trial of labor after cesarean delivery
   4. History of postpartum hemorrhage
   5. ≥4 previous vaginal deliveries
   6. Multiple gestation
   7. The presence of > 2 uterine fibroids or fibroid > 5 cm on any ultrasound during the pregnancy
   8. Planned magnesium sulfate use
   9. Placenta previa/accreta/increta/percreta

Exclusion Criteria:

1. Receipt of anticoagulation (prophylactic anticoagulation stopped 24 hours prior to sample collection is not an exclusion)
2. Antepartum hemorrhage present on admission (>500cc Estimated Blood Loss (EBL))
3. Coagulation defects
4. Thrombocytopenia with platelets count <100,000
5. Enrolled in the "Tranexamic Acid for the Prevention of Obstetrical Hemorrhage After Cesarean (TXA)" (NCT03364491) study or planned receipt of Tranexamic Acid (TXA) prior to enrollment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Pregnant women with high risk of postpartum hemorrhage
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2020-07-27 (Actual); Primary Completion 2021-01-30 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Evaluating degrees of Fibrin polymerization (FIBTEM) ROTEM in the immediate postpartum period. | After delivery through study completion, an average of 2 years

SECONDARY OUTCOMES:
Evaluating INTEM, EXTEM and APTEM Clotting time in pre and post-delivery. | Pre and post-delivery through study completion, an average of 2 years
Evaluating volume of estimated and quantitative blood loss | Pre and post-delivery through study completion, an average of 2 years
Evaluating change in hemoglobin/hematocrit ratio between values on admission for delivery (or in the last 4 weeks prior to delivery) and at 24 (+/-4) hours postpartum | Pre and post-delivery through study completion, an average of 2 years
Evaluating amount of Postpartum hemorrhage defined as Quantitative Blood Loss >500ml for vaginal delivery and >1000ml for cesarean delivery | Pre and post-delivery through study completion, an average of 2 years
Evaluating frequency of blood transfusion and related morbidities | Pre and post-delivery through study completion, an average of 2 years
Evaluating number of severe maternal morbidity (including admission to ICU, intubation, shock) | Pre and post-delivery through study completion, an average of 2 years
Evaluating incidence of need for surgical and non-surgical interventions to manage Postpartum hemorrhage (PPH) | Pre and post-delivery through study completion, an average of 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- The Ohio State University Wexner Medical Center OB/GYN Maternal and Fetal Medicine, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No